CLINICAL TRIAL: NCT06346340
Title: A Phase 4, Multicenter, Open-Label Study to Evaluate the Effect of Miebo™ on Preoperative Biometry/ Keratometry and Postoperative Refractive Accuracy
Brief Title: A Study to Evaluate the Effect of Miebo™ on Preoperative Biometry/Keratometry and Postoperative Refractive Accuracy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 936
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — perfluorohexyl-octan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Miebo treatment (Experimental)
  Interventions: Drug: Miebo

INTERVENTIONS:
Drug: Miebo — Miebo applied in both eyes 4 times per day for approximately 30 days before cataract surgery. Following the completion of the standard follow up, approximately 30 days after cataract surgery, subjects will begin a second regimen of Miebo , 4 times per day in both eyes, for approximately 30 days.

SUMMARY:
A Phase 4, Multicenter, Open-Label Study to Evaluate the Effect of Miebo™ on Preoperative Biometry/ Keratometry and Postoperative Refractive Accuracy

DETAILED DESCRIPTION:
The primary objective is to determine the effect of preoperative Miebo treatment on the accuracy of preoperative biometry/keratometry and predicted refraction in subjects with dry eye disease (DED) who are already scheduled for cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of consent
2. Able to provide written voluntary informed consent
3. The same eye must satisfy the below inclusion criteria (a-e):

   1. At least 1 eye with a visually significant cataract that has been scheduled for cataract surgery (eligible eye can be a subject's second eye to undergo cataract surgery as long as all eligibility criteria are met in that eye)
   2. Candidate for routine, uncomplicated cataract surgery (phacoemulsification with posterior chamber intraocular lens [IOL] implantation, not combined with any other surgery)
   3. In the Investigator's opinion, subject has potential postoperative pinhole Snellen visual acuity of at least 20/200 in both eyes
   4. Tear film break-up time ≤10 sec at Visit 1
   5. Total CFS score ≥2 and ≤11 (ie, sum of inferior, superior, central, nasal, and temporal), using the National Eye Institute scale at Visit 1
4. Ocular Surface Disease Index (OSDI) ≥23 at Visit 1
5. Able and willing to follow instructions, including participation in all trial assessments and visits.

Exclusion Criteria:

1. Have any clinically significant ocular surface slit-lamp findings in the study eye and/or, in the opinion of the Investigator, have any findings that could interfere with trial parameters, including:

   1. History of eye trauma
   2. History of Stevens-Johnson syndrome
   3. Active blepharitis or lid margin inflammation
   4. DED secondary to scarring, irradiation, alkali burns, cicatricial pemphigoid, or destruction of conjunctival goblet cells (as with vitamin A deficiency)
   5. Abnormal lid anatomy causing incomplete eyelid closure
   6. Abnormal cornea shape (keratoconus)
   7. Corneal epithelial defect or significant confluent staining or filaments
   8. History of herpetic keratitis
   9. Ocular or periocular rosacea
2. Pterygium in either eye
3. Use of any of the following ocular therapies in the study eye within 30 days prior to Visit 1: Vuity®, Qlosi™, topical ocular steroid treatments, prescription dry eye therapy including varenicline nasal spray, or topical anti-glaucoma medication
4. Had a LipiFlow® procedure, intense pulse light procedure, or any kind of other procedure affecting meibomian glands in the study eye within 3 months prior to Visit 1
5. Had received or removed a permanent punctum plug in the study eye within 1 month (3 months for dissolvable punctum plugs) prior to Visit 1
6. Use of any eye drops (prescription or over-the-counter, such as artificial tears or Lumify®) and/orTrueTear™ device (intranasal tear neurostimulator) in the study eye within 24 hours prior to Visit 1
7. Have active ocular allergies or ocular allergies that are expected to be active during the trial period
8. Have worn contact lenses within 1 month prior to Visit 1 or planned wear during the study
9. Have undergone intraocular surgery or ocular laser surgery in the study eye within 3 months prior to Visit 1; have undergone refractive surgery in the study eye within 2 years prior to Visit 1
10. Have active ocular or systemic infection (bacterial, viral, or fungal), including fever
11. Female subjects who are pregnant, nursing, or planning a pregnancy
12. Female subjects of childbearing potential who are not using an acceptable means of birth control; acceptable methods of contraception include hormonal (oral, implantable, injectable, or transdermal) contraception; mechanical (spermicide in conjunction with a barrier such as a diaphragm or condom) contraception; intrauterine device; or surgical sterilization of partner. For non-sexually active female subjects, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the trial, she must agree to use adequate birth control as defined above for the remainder of the trial.
13. Have an uncontrolled systemic disease that, in the opinion of the Investigator, will interfere with the trial
14. Have a known allergy and/or sensitivity to the investigational drug
15. Use of any oral medications known to cause ocular drying (eg, antihistamines, antidepressants, etc.) on a non-stable regimen within 1 month prior to Visit 1 or is expected to be unstable during the trial
16. Have taken isotretinoin (eg, Accutane, Myorisan, Claravis, Amnesteem) within 6 months prior to Visit 1
17. Are currently enrolled in an investigational drug or device study or had used an investigational drug or device within 60 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Mean difference between absolute deviations from predicted refractive error in the study eye. | Assessed at Postop Day 30 ± 7 days
  Mean difference between absolute deviations from predicted refractive error in the study eye at Visit 3 (Second Eye/Unilateral Postop Day 30 ± 7 days).

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Site 105, Laguna Hills, California
  - Site 102, Petaluma, California
  - Site 109, Sacramento, California
  - Site 111, Grand Junction, Colorado
  - Site 103, Largo, Florida
  - Site 106, Oak Lawn, Illinois
  - Site 108, Alexandria, Minnesota
  - Site 104, St Louis, Missouri
  - Site 101, Somersworth, New Hampshire
  - Site 107, Sioux Falls, South Dakota
  - Site 110, San Antonio, Texas
  - Site 112, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovanesian JA, Liang E, Desai NR, Berdy GJ, Karpuk K, Schweitzer J, Alexander A, Vittitow JL, Berdahl J, Bacharach J. Perfluorohexyloctane Ophthalmic Solution in Patients with Dry Eye Disease Undergoing Cataract Surgery: A Prospective Multicenter Study. Ophthalmol Ther. 2026 Jan 26. doi: 10.1007/s40123-025-01302-z. Online ahead of print. PMID 41588216